CLINICAL TRIAL: NCT03799809
Title: Efficacy of Intrabronchial Voriconazole Instillation for Inoperable Pulmonary Aspergilloma- a Randomized Controlled Trial
Brief Title: Efficacy of Intrabronchial Voriconazole Instillation for Inoperable Pulmonary Aspergilloma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, DR SACHIN D, senior resident, All India Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS SACHIN
Record Dates: First submitted 2018-10-20; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Aspergilloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voriconazole (Active Comparator): Will receive 400 mg of Intrabronchial Voriconazole every week for 4 weeks along with standard medical therapy.
  Interventions: Drug: Intrabronchial Voriconazole instillation
- Control (No Intervention): Will receive standard medical therapy alone (hemostatics, anti-tussive and others as deemed appropriate by treating physician)

INTERVENTIONS:
Drug: Intrabronchial Voriconazole instillation — Efficacy of intrabronchial voriconazole instillation for inoperable pulmonary aspergilloma
  Arms: Voriconazole

SUMMARY:
Pulmonary aspergillomas are a common cause of recurrent hemoptysis which may be moderate to severe in 2 to 50 % of cases and may be life threatening. Surgical resection, though curative, may not be feasible in significant number of patients and also associated significant post op complications. Bronchial artery embolisation (BAE) is effective for acute control of hemoptysis, however recurrences may occur in upto a quarter of subjects over a 1 year period.

Aspergilloma is caused by a fungus hence systemic antifungals seem appropriate choice. However the fungus only partially touch the walls of the cavities containing them and rarely come into contact with the bloodstream. This is the major reason why the systemic administration of antifungal agents is ineffective in eradicating the condition.

If surgical resection is not a treatment option to control recurrent hemoptysis, instillation of antifungal agents in an aspergilloma cavity could be considered(QoE II).The instillation of antifungal directly into the cavity (intra-cavitatory) containing aspergilloma brings the drug in contact with the fungus. Thus may lead to antifungal action and shrinkage or complete disappearance of aspergilloma. This can be achieved either by percutaneous route or bronchoscopically. Percutaneous approaches have been investigated however they can sometimes cause fungal spread in thoracic space resulting in fungal empyema which should be carefully avoided. Endobronchial instillation of antifungals have been investigated and found to be safe and effective in controlling hemoptysis, however published data comprise of case reports or small case series.

Recently we have published our experience of intrabronchial voriconazole in aspergilloma among 82 patients and found to be safe and effective in hemoptysis control, with transient post procedure cough as an adverse effect with no major serious adverse events. Multiple small studies and case reports have published the safety and efficacy of voriconazole. However, a quality data in the form of randomized controlled trial (RCT) is not there. Therefore, we planned this RCT to assess the efficacy of intrabronchial voriconazole in inoperable aspergilloma.

DETAILED DESCRIPTION:
Primary Objective : To compare the percentage of patients achieving reduction in hemoptysis in intrabronchial voriconazole with standard medical therapy group vs standard medical therapy alone for inoperable symptomatic pulmonary aspergilloma.

Secondary Objectives:

1. To compare the percentage of patients who have complete cessation of hemoptysis after 3 months.
2. To compare the percentage of patients having recurrence of hemoptysis during 3 months follow up.
3. To compare the severity of hemoptysis during recurrence in both groups.
4. To compare the change in size of aspergilloma after 3 - 6 months following last intrabronchial voriconazole instillation.
5. To compare the percentage of patients who need BAE during anytime till 3 - 6months.
6. To compare the percentage of patients with symptomatic improvement in Dyspnea On Exertion, Cough and recurrent respiratory infections.

Number of Patients: 30 patients in each arm (Intrabronchial voriconazole with Standard medical therapy vs Standard medical therapy alone)

Study Design : Prospective Randomized control study

Dosages of drug - 400 mg iv preparation of Voriconazole every week for 4 sessions

Duration of follow-up - 3-6 months

Brief Methodology: Patients with aspergilloma who presented with hemoptysis will be screened for inclusion in the study. Diagnosis of aspergilloma will be based on characteristic computed tomography (CT) features with microbiological or serological evidence of Aspergillus (Aspergillus specific Ig G). The patients fulfilling the inclusion criteria will be taken informed consent and randomized into one of the two arms of intervention.

Arm 1: Will receive 400 mg of Intrabronchial Voriconazole every week for 4 weeks along with standard medical therapy.

Arm 2: Will receive standard medical therapy alone (hemostatics, anti-tussive and others as deemed appropriate by treating physician)

All subjects in arm 1 will undergo fiberoptic bronchoscopy (FOB) following standard protocol under local anesthesia with supplemental oxygen and continuous hemodynamic monitoring. After identifying the segmental/sub-segmental bronchus of interest (as identified by CT) or cavity (if visible) the study drug voriconazole, will be instilled. The bronchoscope will be kept wedged for 60 seconds to prevent back leakage of the solution and then slowly withdrawn without applying suction. The patient will be kept in right or left lateral position (depending on the side of involvement) for the next 20 minutes. Following this patients will be observed for 48 hours for cessation of hemoptysis before discharge. The procedure will be done on day 1 of each week for 4 weeks in arm 1.

All patients will receive standard medical treatment for hemoptysis including appropriate positioning, airway protection, blood product transfusions, antitussives, tranexamic acid, and antimicrobial therapy as clinically indicated. BAE shall be offered to all patients if indicated.

Mild hemoptysis shall be defined as < 50 ml in 24 hrs, moderate hemoptysis as 50-200 ml in 24 hrs and massive hemoptysis as 200-600 ml in 24 hrs or any amount causing hemodynamic compromise/threatening ventilation.

Records will be reviewed regarding demographics, primary etiology leading to fibrocavitary disease, duration and severity of hemoptysis/ other constitutional symptoms, extent of disease (unilateral, bilateral, associated pleural or parenchymal changes), simple vs complex aspergilloma. Size of index aspergilloma. The number of patients requiring emergency or hospital admission due to recurrent hemoptysis, and subsequent treatment details will be recorded.

All patients will be followed up for 3-6 months. During follow up patients will be assessed for symptoms and severity, successful cessation of hemoptysis, requirement of BAE due to persistent or increased hemoptysis, number of sessions required for symptomatic improvement/cessation of hemoptysis, hemoptysis-free interval, recurrence of hemoptysis will be noted. Pre and post procedure CT scans (low dose limited CT through aspergilloma) will be compared by an independent radiologist blinded to the clinical outcome. Size of index aspergilloma shall be determined by addition of maximum diameter of largest length and width of the visible lesion. CTs shall be compared for documenting change in the size of index aspergilloma and decrease/disappearance of the cavity. On the basis of these parameters, aspergillomas will be described as no interval change, increased or decreased aspergilloma size, or disappearance and emptying of the cavity.

Outcomes in the form of reduction/cessation of hemoptysis, decrease in size of aspergilloma, overall symptomatic improvement and mortality shall be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate hemoptysis AND inoperable aspergilloma/ those unwilling for surgery.
* Who have no contra-indication of flexible fibre-optic bronchoscopy
* Age > 18 yrs AND
* Given the written informed consent to participate in the study.

Exclusion Criteria:

* Patient who are not fit for FOB (e.g. hemodynamic instability)
* Patient who have life threatening hemoptysis requiring immediate bronchial artery embolization
* Patients who have underwent BAE in last 3 months
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
To compare the percentage of patients achieving reduction in hemoptysis in intrabronchial voriconazole with standard medical therapy group vs standard medical therapy alone for inoperable pulmonary aspergilloma at 3 months. | 3 months follow up
  Percentage of patients achieving reduction in hemoptysis in intrabronchial voriconazole with standard medical therapy group vs standard medical therapy alone for inoperable pulmonary aspergilloma at 3 months.

SECONDARY OUTCOMES:
To compare the percentage of patients who have complete cessation of hemoptysis after 3 months. | 3 months follow up
  percentage of patients who have complete cessation of hemoptysis after 3 months.
To compare the percentage of patients having recurrence of hemoptysis during 3 months follow up. | 3 months follow up
  percentage of patients having recurrence of hemoptysis during 3 months follow up.
To compare the severity of hemoptysis during recurrence in both groups. | 3 months follow up
  severity of hemoptysis during recurrence in both groups shall be compared with visual analogue scale.
To compare the change in size of aspergilloma after 3 months following last intrabronchial voriconazole instillation. | 3 months follow up
  change in size of aspergilloma after 3 months following last intrabronchial voriconazole instillation.
To compare the percentage of patients who need BAE during anytime till 3 months. | 3 months follow up
  percentage of patients who need BAE during anytime till 3 months.
To compare the percentage of patients with symptomatic improvement in Dyspnea On Exertion, Cough and hemoptysis. | 3 months follow up
  percentage of patients with symptomatic improvement in Dyspnea On Exertion, Cough and hemoptysis.

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No